CLINICAL TRIAL: NCT00665704
Title: Tobacco Tactics Website for Veteran Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SHP 08-197
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-06

CONDITIONS: Smoking
Keywords: Smoking Cessation; Internet; Intervention Studies; Health Services Accessibility
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tobacco Tactics Website (Experimental): Nine veteran smokers who will pilot test the Tobacco Tactics website
  Interventions: Behavioral: Tobacco Tactics website

INTERVENTIONS:
Behavioral: Tobacco Tactics website — Pilot test the Tobacco Tactics website tailored to the needs of veteran smokers

SUMMARY:
The purpose of this study is to develop an evidence-based Tobacco Tactics website tailored to veterans based on an intervention tested in the VA.

DETAILED DESCRIPTION:
Despite the detrimental effects of smoking, approximately 33% of veterans continue to smoke compared to approximately 21% of the general population. While efficacious cessation interventions are available, implementation of cessation interventions remains a challenge and new intervention strategies are needed to reach veterans. VA cessation providers recently met in Atlanta and one recommendation was to develop a cessation website for veterans. The evidence-based Tobacco Tactics website will be designed, pre-tested, and pilot tested as an intervention to assist veteran smokers to quit smoking. The efficacy of the website will then be tested in a subsequent randomized control trial (RCT). If the website proves efficacious, it would decrease morbidity and mortality among veterans, decrease face-to-face cessation intervention time for providers, and reach veterans in areas all over the country, perhaps through the VA "My Healthy Vet" website. This is a Phase 1 behavioral clinical trial designed to develop and pilot test a web-based Tobacco Tactics intervention tailored to veteran smokers. First, we will outline the specific content areas to be addressed. Second, we will develop the Tobacco Tactics intervention with our web designer in accordance with VA Web Operations. Third, a member of the research team will go through the website with the 5 veteran smokers obtaining feedback and noting any problems that occur. Fourth, with human studies approval, we will pilot test the impact of the intervention with 9 veteran smokers recruited to quit smoking using the Tobacco Tactics website. A research nurse will:

1. be available by phone to answer any questions;
2. collect qualitative data on veterans use of the Tobacco Tactics website; and,
3. note the 30 day quit rate.

Formative evaluation during pre-testing will include qualitative feedback on the:

1. ability to accomplish tasks;
2. ability to accomplish goals with skill and speed;
3. ability to operate the system; and
4. satisfaction.

For the 9 veteran smokers that actually try to use the Tobacco Tactics website to quit smoking, we will be able to determine:

1. the number of times they signed onto the website;
2. the time spent on the website; and
3. the number of times each module was accessed.

Impact evaluation will be the 30 day quit rates of the 9 veteran smokers that agree to use the website.

ELIGIBILITY:
Inclusion Criteria:

* Veteran,
* Screen Positive for Current Smoking,
* Greater than 18 Years of Age,
* Access to the Internet

Exclusion Criteria:

* Non-English Speaking,
* Have Unstable Physical or Psychiatric/Mental Conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia A. Duffy, PhD MS RN, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Duffy SA, Fowler KE, Flanagan PS, Ronis DL, Ewing LA, Waltje AH. The development of the tobacco tactics website. JMIR Res Protoc. 2013 Jun 28;2(2):e22. doi: 10.2196/resprot.2445. PMID 23811612

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tobacco Tactics Website
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tobacco Tactics Website
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 48 [29 to 63]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Self Reported 30 Day Smoking Quit Rate
Description: Impact evaluation was the 30-day quit rates of the 9 veteran smokers that agreed to use the website.
Time Frame: 30 days post intervention
Measure: Number; unit: participants
Arm/Group | Tobacco Tactics Website
Number analyzed (Participants) | 9
participants | 0

2. Secondary Outcome: Patient Feedback to Evaluate the Website
Description: Formative evaluation during pre-testing included qualitative feedback on the: 1) ability to accomplish tasks; 2) ability to accomplish goals with skill and speed; 3) ability to operate the system; and 4) satisfaction. For the 9 veteran smokers that actually tried to use the Tobacco Tactics website to quit smoking, we were able to determine: 1) the number of times they signed onto the website; 2) the time spent on the website; and 3) the number of times each module was accessed.
Time Frame: 30 days post intervention
Measure: Number; unit: participants
Arm/Group | Tobacco Tactics Website
Number analyzed (Participants) | 9
participants
  easy to read | 5
  enjoyable | 4
  easy to navigate | 4

ADVERSE EVENTS:
Arm/Group | Tobacco Tactics Website
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No